CLINICAL TRIAL: NCT06033170
Title: Prospective, Single-Arm Confirmatory Clinical Investigation to Demonstrate the Effectiveness, Performance, and Safety of the Celox™ PPH for Reaching Haemostasis in Patients With Postpartum Hemorrhage
Brief Title: Celox™ PPH for Reaching Haemostasis in Patients With Postpartum Hemorrhage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medtrade (Industry)
Collaborators: Charite University, Berlin, Germany (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PMCF_PPH 01
Record Dates: First submitted 2023-07-25; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Insertion of CELOX™ PPH trans-vaginally for bleeding control (Experimental): There is only one group.
  Interventions: Device: CELOX™ PPH

INTERVENTIONS:
Device: CELOX™ PPH — Celox™ PPH is intended to be a physical haemostatic treatment for control and treatment of uterine postpartum hemorrhage (PPH) when conservative management is warranted.

SUMMARY:
This is a post market prospective, single arm clinical investigation to continuously assess the safety performance and effectiveness of the Celox™ PPH as a uterine haemostatic tamponade treatment for uterine postpartum hemorrhage (PPH).

ELIGIBILITY:
Inclusion Criteria:

* Subject or her legally authorized representative is able to understand and provide consent to participate in the clinical investigation
* Female Adult subjects (>18 years of age).
* Diagnosis of PPH with suspected uterine atony placental bed bleeding, placenta accreta or previa within 24 hours after vaginal delivery.
* Subjects with coagulation disorders can be included
* Minimal Estimated Blood Loss (EBL), to be determined when investigator is ready to have the Celox™ PPH package opened. 500 ml of EBL for vaginal delivery or 1000 ml for caesarean section.
* Failed first-line intervention of uterotonics and uterine massage/bimanual compression to stop bleeding. Note: Uterotonic administration may continue concomitant with and post the Celox™ PPH use.
* Subjects with PPH of cervical or vaginal origin.

Exclusion Criteria:

Subjects who present with, uterine rupture or for any other conditions outside of atonic post-partum haemorrhage needing other interventional methods or surgery including uterine artery embolization (UAE).

* Pregnancy or incomplete multiple pregnancy
* Unresolved uterine inversion.
* Current cervical cancer.
* Current purulent infection of the vagina, cervix, uterus.
* Planned c-section with closed cervix.
* Patients requiring trans-abdominal insertion of Celox™ PPH.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Celox™ PPH in controlling uterine bleeding in postpartum hemorrhage (PPH). | Successful haemostasis is defined as absence of additional surgical or non-surgical interventions after application of Celox PPH. It is expected that within 2-5 minutes of application, the bleeding will be controlled.
  The rate of patients in whom bleeding is controlled successfully.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Maria Dückelmann, MD, Principal Investigator — Charite University, Berlin, Germany; NIK Abdullah, MD, Principal Investigator — Hospital Raja Perempuan Zainab II - Malaysia

IPD SHARING:
Plan to Share IPD: No